CLINICAL TRIAL: NCT04091620
Title: Transanal Total Mesorectal Excision Versus Robotic Total Mesorectal Excision for Mid and Low Rectal Cancer: A Prospective Randomized Controlled Trial
Brief Title: Transanal Total Mesorectal Excision Versus Robotic Total Mesorectal Excision
Acronym: TaRo
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Simon S. M. Ng, Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CREC 2019.072
Record Dates: First submitted 2019-09-14; First posted 2019-09-17 (Actual); Last update posted 2019-10-04 (Actual); Status verified 2019-09

CONDITIONS: Rectal Cancer
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Transanal Total Mesorectal Excision (Experimental): For transanal total mesorectal excision, a two team approach will be adopted. One surgical team will be performing the abdominal phase dissection using standard laparoscopic approach, while the other will be simultaneously performing the transanal dissection and total mesorectal excision in a 'down-to-up' fashion using laparoscopic instruments.
  Interventions: Procedure: Transanal Total Mesorectal Excision
- Robotic Total Mesorectal Excision (Active Comparator): For robotic total mesorectal excision, a fully robotic approach will be adopted. Left-sided colonic mobilization, division of lymphovascular pedicle, and 'top-to-down' total mesorectal excision will be performed using the robotic platform.
  Interventions: Procedure: Robotic Total Mesorectal Excision

INTERVENTIONS:
Procedure: Transanal Total Mesorectal Excision — As above
  Arms: Transanal Total Mesorectal Excision
Procedure: Robotic Total Mesorectal Excision — As above
  Arms: Robotic Total Mesorectal Excision

SUMMARY:
Background: Laparoscopic total mesorectal excision (TME) for rectal cancer is technically challenging because of the confined space within the pelvis. The robotic surgical system is recently introduced to overcome the limitations of laparoscopy in terms of visualization and maneuverability, but robotic surgery is expensive. Transanal total mesorectal excision (TaTME) is an emerging surgical approach that allows dissection of the most difficult part of the TME plane deep down in the pelvis using a less costly transanal platform. To date, no randomized controlled trial can be found in the literature comparing TaTME and robotic TME.

Objectives: To compare the pathologic outcomes, functional outcomes, and costs between TaTME and robotic TME for mid or low rectal cancer.

Design: Prospective, randomized, controlled, superiority trial.

Subjects: One hundred and eight consecutive patients who are clinically diagnosed with cT1-3, N0-2, M0 rectal cancer located within 12 cm of the anal verge who do not require abdominoperineal resection will be recruited.

Interventions: Patients will be randomly allocated to undergo either TaTME or robotic TME.

Outcome measures: Primary outcome: composite pathologic endpoint (complete TME, clear circumferential and distal resection margins). Secondary outcomes: conversion rate, postoperative recovery, morbidity, health-related quality of life, urosexual function, and costs.

Hypothesis: Results of the present study can provide evidence-based clarification of the efficacy and safety of TaTME for patients with mid and low rectal cancer. The results of this proposed project may have a significant impact on the future treatment strategy for mid and low rectal cancer.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive patients who are diagnosed with mid or low rectal adenocarcinoma, of which the lowest margin of the tumor is located at or within 12 cm of the anal verge as determined by rigid sigmoidoscopy
* Those with clinically diagnosed cT1-3, N0-2, M0 disease based on preoperative staging with pelvic magnetic resonance imaging, computed tomography, and/or positron emission tomography
* Age of patients greater than or equal to 18 years
* Those with American Society of Anesthesiologists (ASA) grading I-III,
* Informed consent available

Exclusion Criteria:

* Patients with locally advanced cancer not amenable to curative surgery (e.g. involved mesorectal fascia on pelvic magnetic imaging despite neoadjuvant chemoradiotherapy)
* Those with locally advanced T4 cancer requiring en bloc multivisceral resection
* Those with very low rectal tumor requiring abdominoperineal resection
* Those with synchronous colorectal tumors requiring multisegment resection
* Those undergoing emergency surgery
* Those with previous history of abdominal surgery precluding the robotic or laparoscopic approach;
* Those with severe cardiopulmonary disease rendering pneumoperitoneum hazardous
* Those with psychiatric disease
* Those who are pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2019-10-01 (Actual); Primary Completion 2022-10 (Estimated); Study Completion 2022-10 (Estimated)

PRIMARY OUTCOMES:
Incidence rate of achieving a composite of pathologic endpoint indicating adequate surgical resection | Up to 1 month
  Achieving a composite pathologic endpoint or a successful resection is defined as meeting all the following criteria: (1) complete total mesorectal excision, (2) clear circumferential resection margin (>1 mm), and (3) clear distal resection margin (> 1mm).

SECONDARY OUTCOMES:
Rate of conversion | Up to 1 month
  Conversion is defined as an abdominal incision larger than necessary for specimen retrieval for the abdominal phase of transanal total mesorectal excision (TME) and robotic TME; for the transanal phase of transanal TME conversion is defined as failure to complete a 'down-to-up' TME transanally, and the majority of the TME has to be completed using the abdominal approach.
Time to defecation | Up to 1 month
Time to resume full solid diet | Up to 1 month
Time to walk independently | Up to 1 month
Length of hospital stay | Up to 1 month
Pain scores on visual analog scale | Up to 1 month
  From 0 which implies no pain at all, to 100 which implies the worst pain imaginable, on the first 3 postoperative days.
Morbidity within 30 days | Up to 1 month
  Surgical complications are classified according to the Clavien-Dindo classification.
Urinary function at 3, 6, 9, and 12 months after surgery, measured by the International Prostate Symptom Score (IPSS) | Up to 12 months
  IPSS is based on the answers to seven questions concerning urinary symptoms and one question concerning quality of life. Each question concerning urinary symptoms allows the patient to choose one out of six answers indicating increasing severity of the particular symptom. The answers are assigned points from 0 to 5. The total score can therefore range from 0 to 35 (asymptomatic to very symptomatic).
Male sexual function at 3, 6, 9, and 12 months after surgery, measured by the International Index of Erectile Dysfunction - 5 (IIEF-5 questionnaire) | Up to 12 months
  IIEF-5 is an abridged five-item version of the 15-item International Index of Erectile Function (IIEF) which is used to diagnose the presence and severity of erectile dysfunction. This questionnaire consists of only five questions and each IIEF-5 item is scored on a five-point ordinal scale where lower values represent poorer sexual function. Thus, a response of 0 for a question is considered the least functional, whereas a response of 5 is considered the most functional. The possible scores for the IIEF-5 range from 1 to 25 (one question has scores of 1-5), and a score above 21 is considered as normal erectile function and at or below this cutoff, erectile dysfunction.
Anal continence at 3, 6, 9, 12 months after surgery, measured by the Cleveland Clinic Incontinence Score (Wexner's Score) | Up to 12 months
  The Cleveland Clinic Incontinence Score or Wexner's Score is the most common score used to determine the severity of incontinence before and after surgery for anal incontinence. The scoring system takes into account the type and frequency of incontinence, and the extent to which it alters the patient's life. It consists of five questions to assess the degree of incontinence (solid, liquid, gas, wears pad, lifestyle alteration). The frequency of each type of incontinence is rated on a scale ranging from 0 (never) to 4 (always or to once a day) so that the sum of the frequencies add up to a total score that may range from 0 to 20. Higher scores indicate higher levels of incontinence.
Quality of life scores measured by Short Form 36 (SF-36) Health Survey at 3, 6, 9, 12 months after surgery | Up to 12 months
  The Short Form 36 (SF-36) Health Survey is a 36-item, patient-reported survey of patient health. It consists of eight scaled scores, which are the weighted sums of the questions in their section. The eight sections are: vitality, physical functioning, bodily pain, general health perceptions, physical role functioning, emotional role functioning, social role functioning, and mental health. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability i.e., a score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability.
Quality of life scores measured by European Organisation for Research and Treatment of Cancer (EORTC) QLQ-C30 questionnaires at 3, 6, 9, 12 months after surgery | Up to 12 months
  EORTC QLQ-C30 is a generic questionnaire for assessment of quality of life (QoL) in cancer patients. It includes 30 items, 24 of which are combined to form a global QoL scale, five functional scales (physical, role, emotional, cognitive, and social), and three symptom scales (fatigue, nausea/vomiting, and pain). The other six single items evaluate dyspnea, insomnia, appetite loss, constipation, diarrhea, and financial difficulties. All questionnaires responses and scores will be linearly transformed to a 0-100 scale. A higher score on the global QoL and functional scales represents a higher level of QoL and functioning, whereas a higher score on the symptom scales/items represents a higher degree of symptoms or dysfunction.
Quality of life measured by European Organisation for Research and Treatment of Cancer (EORTC) QLQ-CR38 questionnaires at 3, 6, 9, 12 months after surgery | Up to 12 months
  EORTC QLQ-CR38 is a specific questionnaire module specifically designed for assessment of quality of life (QoL) in patients with colorectal cancer. It consists of 38 items covering symptoms and side effects related to different colorectal cancer treatment modalities. The module contains four functional scales (body image, sexual functioning, sexual enjoyment, and future perspective) and eight symptom scales/items (micturition problems, chemotherapy side effects, gastrointestinal tract symptoms, male sexual problems, female sexual problems, defecation problems, stoma-related problems, and weight loss). All questionnaires responses and scores will be linearly transformed to a 0-100 scale. A higher score on the global QoL and functional scales represents a higher level of QoL and functioning, whereas a higher score on the symptom scales/items represents a higher degree of symptoms or dysfunction.
Direct/indirect medical costs and out-of-hospital economic costs | Up to 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Simon SM Ng, MD, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Prince of Wales Hospital, The Chinese University of Hong Kong, Hong Kong, China

IPD SHARING:
Plan to Share IPD: No